CLINICAL TRIAL: NCT07175454
Title: A Study to Describe the Burden of Mental Ill Health in Inflammatory Bowel Disease Patients Using Advanced Therapies, and to Identify Any Associations Between Common Mental Health Problems and the Efficacy of Such Advanced Therapies (IBDmind)
Brief Title: IBDminds - Mapping the Influence of aNxiety and DepreSsion on IBD
Acronym: IBDminds
Status: Not yet recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025GAS146
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Diseases; Mental Health Issue
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Patients/research nurses will complete questionnaires detailing their medical history including mental health and describing their IBD.
  Patients will complete baseline scoring questionnaires for depression and anxiety (HADS) and perceived stress (PSS-10).
  Patients will also complete a patient reported outcome tool to assess their current disease activity level (PRO-2)

SUMMARY:
People with Inflammatory bowel disease (IBD) can get challenging symptoms. Things like diarrhoea, tummy pain and being tired all the time are common. People often get IBD in their teens or twenties. They often find working, studying and relationships hard. IBD can't be cured, so it lasts for life.

When IBD is hard to treat, we use advanced treatments, but these don't always work. When they do work the effect can wear off. This happens in 2 of 5 people within a year in research studies. There are some things that we know make them wear off. There are lots more reasons that we don't understand yet. We think anxiety, depression and stress make these treatments more likely to wear off. Previous research has suggested that people with IBD do worse if they have anxiety, depression or stress.

The investigators want people with IBD to complete questionnaires to see if they are affected by anxiety, depression or stress when they are taking advanced therapies. The investigators will follow those people to see if the effect of their treatment wears off.

People living with IBD will contribute to the running and fine tuning of this research. Many of those that have engaged with us so far have said that their disease was worse when their mental health was worse. They were generally supportive of this study to see how anxiety, depression and stress effects IBD in people using advanced therapies.

The investigators have talked to a national charity about our work. They will help share the findings so that patients, care givers and other stakeholders will be able to read about them. The results will be published so that doctors and researchers can use them.

DETAILED DESCRIPTION:
The treatment of moderate to severe Inflammatory Bowel Disease (IBD) now consists of a wide selection advanced therapies1. Despite these, the efficacy of advanced therapy has reached a ceiling at approximately 40% of patients achieving remission. Furthermore, a significant proportion will lose response to the medication within 1 year of starting2-4, which is likely to be multi-factorial.

There is a recognised association between IBD and common mental health problems, specifically anxiety, depression and perceived stress, but it is not known whether these impact the effectiveness of IBD treatment.

The bidirectional relationship between mental wellbeing and IBD has been described in a recent meta-analysis5. Patients with anxiety and depression are more likely to develop IBD compared to matched controls without IBD6. This relationship predates IBD presentation by up to 5 years. Therefore, it appears that a complex relationship between IBD and anxiety, depression and perceived stress exists. IBD patients with concurrent anxiety, depression and perceived stress are more likely to have more severe IBD, including; exacerbations, hospital admissions, and need for surgery5.

High levels of perceived personal stress are associated with increased risk of disease exacerbations7. A single study from 2005 demonstrated worse IBD outcomes in patients with severe depression compared to mentally well patients when treated with a single dose of Infliximab (albeit in a practice which is now obsolete). This suggests severe depression is associated with worse outcomes from advanced therapies but further research is needed to validate this association8.

Data to describe a relationship between IBD and anxiety, depression and perceived stress, in patients on advanced therapies is limited. Up to 20% of IBD patients are now progressing to advanced therapies compared to 5% in 20109. Such data is important to consider if intervention for anxiety, depression and perceived stress could improve durability of advanced therapies.

Public contributors to research have articulated that mental health is a key concern. It is a common lived experience amongst patients with IBD that anxiety, depression and perceived stress are a factor in their disease activity. The investigators hypothesise that unrecognised or inadequately managed anxiety, depression and perceived stress is a factor that makes advanced therapies less effective in maintaining remission for IBD patients.

There are also important health inequality considerations. IBD Patients are more likely to develop anxiety and depression if they are from a deprived background, but are also more likely to have worse outcomes from IBD because of anxiety and depression. Worse IBD leads to greater challenge in the workplace and therefore risk of unemployment and increasing deprivation. Research that defines and reduces the negative impact of anxiety and depression on IBD outcomes would also reduce inequality of outcomes driven by deprivation.

The burden of anxiety and depression is increasing10. Current incidence rates amongst any IBD patient using primary care coded data suggest that the incidence of anxiety and depression are 5.5 and 11 per 1000 patient years11. The prevalence of depression at diagnosis has been reported to be 7%6. However, a survey of Australian IBD patients using a combined measure of depression and anxiety found that 50% of patients reported symptoms12. Therefore, the investigators expect a high proportion of patients recruited to this study will report at least some elements of anxiety, depression and perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of ulcerative colitis, or Crohn's disease, based upon either the outcome of the local multidisciplinary team, clinic documentation or in the opinion of the investigator
* Patients receiving maintenance infliximab or vedolizumab by regular intravenous infusion
* Patients willing and able to give informed consent
* Patients aged 16 or over

Exclusion Criteria:

* Patients cannot be recruited while receiving their loading dose of infusions, but may be included once complete.
* Patients should not currently be planned for surgery within the next 12 months
* Patients should not currently be planned to switch to another advanced therapy within the next 12 months
* Patients should not currently be planned for a drug holiday within the next 12 months
* Patients should not have a stoma (This would invalidate the PRO-2 outcome measure)
* Patients should not currently be pregnant
* Patient currently receiving subcutaneous infliximab or vedolizumab

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving IV infliximab or vedolizumab for IBD
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome-2 (PRO-2) | Every 4 weeks over the course of a year
  PRO-2 is an established patient reported outcome measure for IBD. There are separate measurement tools for UC and CD. In UC patients report the rectal bleeding sub-score and stool frequency sub-score from the clinical Mayo score. In CD patients report 3 days of the number of liquid or soft stools and severity of abdominal pain. In both UC and CD the score is well validated to Mayo clinical score and CDAI respectively, and to faecal biomarkers.
Patient Health Questionnaire-9 (PHQ-9) | Every 4 weeks over the course of a year
  PHQ-9 is a self-administered measure of depressive symptoms over the previous 2 weeks. Questions include 9 domains, asking patients to report the frequency of each. PHQ is-9 is mapped to the DSM-4 diagnosis of major depression and therefore offers robust evidence of depression. Although not specifically designed for physical health problems, validity in this group has been demonstrated. PHQ-9 is also sensitive to change, therefore is well suited to serial measurements.
Generalised Anxiety Disorder-7 (GAD-7) | Every 4 weeks over the course of a year
  GAD-7 is a self-administered measure of anxiety over the proceeding 2 weeks. Questions cover 7 domains asking patients to record the frequency of each. GAD-7 is the current UK standard for scale for anxiety utilised in primary care.
Perceived Stress Scale (PSS-10) | Every 4 weeks over the course of a year
  PSS-10 is a self-administered measure of symptoms suggestive of stress over the previous 4 weeks. Questions include ;10 domains, asking patients to report the subjective frequency of each. Stress is an important outcome measure as there is a recognised association with active IBD.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No